CLINICAL TRIAL: NCT01390272
Title: Randomized Trial of Titrated Disease Management for Patients With Hypertension
Brief Title: Titrated Disease Management for Patients With Hypertension
Acronym: TDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 10-383
Record Dates: First submitted 2011-07-06; First posted 2011-07-11 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Hypertension
Keywords: Hypertension; Telephone; Disease Management; Veterans; Pharmacists; Nurses
MeSH Terms: conditions — Hypertension | interventions — Immunization, Secondary; Culture Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titration Intervention (Experimental): The intervention arm includes three levels of resource intensity targeted to improve patients' systolic blood pressure (SBP) [top number of blood pressure measurement].
  Medium/level 1 resource intensity: a registered nurse (RN) will provide monthly tailored behavioral support telephone calls + home BP monitoring.
  High/level 2 resource intensity: a pharmacist will provide monthly tailored behavioral support telephone calls + home BP monitoring + pharmacist-directed medication management.
  Booster (low) resource intensity: a licensed practical nurse (LPN) will provide non-tailored behavioral support telephone calls every two months to patients whose SBP comes under control.
  Interventions: Behavioral: Booster/ low resource; Behavioral: Medium/Level 1 resource intensity; Behavioral: High/Level 2 resource intensity
- LPN Control (Active Comparator): A LPN will provide behavioral support telephone calls that do not include goal setting and directed problem solving every two months (identical to booster (low) resource intensity component of the titrated intervention). The control arm will utilize the same procedures as the booster level for intervention patients for whom SBP comes under control.
  Interventions: Behavioral: Booster/ low resource

INTERVENTIONS:
Behavioral: Booster/ low resource — A LPN will provide behavioral support telephone calls that do not include goal setting and directed problem solving every two months.
  Other Names: Control Arm - Low resource
  Arms: LPN Control
Behavioral: Booster/ low resource — A LPN will provide behavioral support telephone calls that do not include goal setting and directed problem solving every two months.
  Other Names: Intervention Arm - Booster
  Arms: Titration Intervention
Behavioral: Medium/Level 1 resource intensity — Monthly tailored RN delivered calls + home BP monitoring.
  Other Names: Intervention Arm - Level 1
  Arms: Titration Intervention
Behavioral: High/Level 2 resource intensity — Pharmacist delivered telephone behavioral self-management support + Home BP monitoring with feedback to pharmacist + Algorithmic medication changes directed by pharmacist (with physician backup).
  Other Names: Intervention Arm - Level 2
  Arms: Titration Intervention

SUMMARY:
This randomized clinical trial examines whether programs aimed at matching resources to patient hypertension (i.e. high blood pressure) control lead to greater reduction in systolic blood pressure (top number of blood pressure reading) than simply having maintenance phone calls in addition to usual care. Answering this question will provide important evidence concerning the overall goal of sustained long-term implementation of the disease management programs as part of patient aligned care teams in the Veterans Affairs and other healthcare systems.

DETAILED DESCRIPTION:
Project Objectives: The investigators are conducting a two-arm 18-month randomized clinical trial for patients with pharmaceutically treated hypertension for which systolic BP is not controlled (>/=140 mmHg for non-diabetic or >/=130 mmHg for diabetic patients). The primary aim will be to compare two treatment arms/strategies in terms of impact on systolic BP control: Arm 1 - An intervention arm using titrated disease management in which patients' hypertension control, assessed at baseline, 6 and 12 months, will be used to decide the resource intensity of strategies: 1) Medium/level 1 resource intensity strategy: a registered nurse will provide monthly tailored behavioral support telephone calls + home BP monitoring; 2) High/level 2 resource intensity strategy: a pharmacist will provide monthly tailored behavioral support telephone calls + home BP monitoring + pharmacist-directed medication management; and 3) Booster (low) resource intensity strategy: a license practice nurse (LPN) will provide bi-monthly, non-tailored behavioral support telephone calls to patients whose systolic BP comes under control. Arm 2 - A control arm, in which an LPN will provide bi-monthly non-tailored behavioral support telephone calls (same procedures as the booster (low) resource intensity strategy component of the titrated intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Assigned primary care provider in one of the clinics of the Durham VA Medical Center (VAMC) (including Community Based Outpatient Clinics for example - Hillandale Clinic and Greenville (CBOC)).
* Had at least 1 primary care visit at the Durham VA or affiliated CBOC in the last year.
* Diagnosis of hypertension requiring medication, as determined by: ICD 401.0, 401.1, or 401.9 for >= 2 outpatient encounters during the prior year and Received a prescription for at least 1 of the following classes of hypertensive medication in the previous year: 1) ACE inhibitors; 2) alpha blockers; 3) angiogenesis II inhibitors; 4) beta blockers; 5) calcium channel blockers; 6) diuretics; 7) antihypertensive combination; and/or 8) antihypertensives, other.
* Out of control systolic blood pressure: Durham VAMC (including CBOCs or other affiliated clinics captured in the Durham VAMC electronic health record) outpatient BP measurements >= 150 mmHg for non-diabetic or >= 140 mmHg for diabetic patients over the last year and last systolic BP measurement >= 140 mmHg for non-diabetic or >= 130 mmHg for diabetic patients. If additional patients need to be approached to be offered the opportunity for further screening, non-diabetic patients with mean outpatient systolic BP of >= 140 mmHg or diabetic patients with mean outpatient systolic BP of >= 130 mmHg over the past year may be approached.

Patients must indicate that they both:

* Have a VA or affiliated clinic provider that they consider to be their main PCP.
* Receive the majority of healthcare at the Durham VA Medical Center (or affiliated clinic - such as Hillandale or Greenville).

Exclusion Criteria:

* Active diagnosis of psychosis.
* Diagnosis of metastatic cancer.
* Type 1 diabetes
* Class IV congestive heart failure (CHF).
* Currently receiving kidney dialysis or if estimated glomerular filtration rate (eGFR) levels are <= 15.
* Chronic obstructive pulmonary disease (COPD) requiring oxygen.
* Resident in nursing home or receiving home healthcare.
* Patient is pregnant or reports planning to become pregnant in the next two years
* At the time of potential enrollment, participating in another ongoing hypertension, diabetes, cholesterol, or cardiovascular disease clinical trial.
* Planning to leave the area prior to the anticipated end of participation.
* Inability or unwillingness to come to the Durham VAMC or affiliated clinic such as Hillandale or Greenville for baseline-, 6-, 12-, and 18-month study visits.
* Does not have reasonable access to a telephone.
* Does not speak English.
* Severely impaired hearing or speech (Patients must be able to respond to phone calls.).
* Severely impaired vision (Patients must be able to read mailed material).
* Refusal or inability to provide informed consent and HIPAA authorization form.
* Arm size > 50 cm
* Unable to obtain (including by arm) valid blood pressure readings
* Inadequate mental status to complete the protocol, as judged by five or more errors on the Short Portable Mental Status Questionnaire (SPMSQ).
* Former, current or pending solid organ or bone marrow transplant patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2012-07-27 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Jackson, PhD MHA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jackson GL, Weinberger M, Kirshner MA, Stechuchak KM, Melnyk SD, Bosworth HB, Coffman CJ, Neelon B, Van Houtven C, Gentry PW, Morris IJ, Rose CM, Taylor JP, May CL, Han B, Wainwright C, Alkon A, Powell L, Edelman D. Open-label randomized trial of titrated disease management for patients with hypertension: Study design and baseline sample characteristics. Contemp Clin Trials. 2016 Sep;50:5-15. doi: 10.1016/j.cct.2016.07.009. Epub 2016 Jul 12. PMID 27417982
- [Result] Jackson GL, Stechuchak KM, Weinberger M, Bosworth HB, Coffman CJ, Kirshner MA, Edelman D. How Views of the Organization of Primary Care Among Patients with Hypertension Vary by Race or Ethnicity. Mil Med. 2018 Sep 1;183(9-10):e583-e588. doi: 10.1093/milmed/usx111. PMID 29672720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted among patients receiving primary care at the Durham VAMC, including VA Community Based Outpatient Clinics (CBOC).
Groups:
- Titration Intervention: The intervention arm includes three levels of resource intensity targeted to improve patients' systolic blood pressure (SBP) [top number of blood pressure measurement].
  Medium/level 1 resource intensity: a registered nurse (RN) will provide monthly tailored behavioral support telephone calls + home BP monitoring.
  High/level 2 resource intensity: a pharmacist will provide monthly tailored behavioral support telephone calls + home BP monitoring + pharmacist-directed medication management.
  Booster (low) resource intensity: a licensed practical nurse (LPN) will provide non-tailored behavioral support telephone calls every two months to patients whose SBP comes under control.
  Booster/ low resource: A LPN will provide behavioral support telephone calls that do not include goal setting and directed problem solving every two months.
Period: Overall Study
Arm/Group | Titration Intervention | LPN Control
Started | 192 | 193
6 Month Follow up | 162 (30 of 192 participants in the Titration Intervention group had missing blood pressure measurement) | 171 (22 of 193 in the LPN control group had missing blood pressure measurement)
12 Month Follow up | 139 (53 of 192 participants in the Titration Intervention group had missing measurement) | 159 (34 of 193 in the LPN control group had missing blood pressure measurement)
18 Month Follow up | 155 (37 of 192 participants in the Titration Intervention group had missing blood pressure measurement) | 160 (33 of 193 in the LPN control group had missing blood pressure measurement)
Completed | 175 | 178
Not Completed | 17 | 15
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 9 | 5
Not completed — Patient moved, no longer eligible | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Titration Intervention | LPN Control | Total
Number analyzed (Participants) | 192 | 193 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Baseline Visit
  years | 64.2 (9.0) | 62.9 (8.5) | 63.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 176 | 180 | 356

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Continuous change in systolic blood pressure was measured as the primary outcome. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the baseline study visits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 192 | 193
mmHg | 143.5 (17.7) | 143.7 (17.5)

2. Primary Outcome: Systolic Blood Pressure
Description: Continuous change in systolic blood pressure was measured as the primary outcome. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the 6- month study visits.
Time Frame: 6 months
Population: 30 out of the 192 participants in the Titration Intervention group and 22 out of the 193 in the LPN control group had missing blood pressure measurement at 6 months due to not completing the assessment. One additional participant in the LPN control had missing blood pressure measurement at 6 months due to not being able to get a reading.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 162 | 171
mmHg | 137.1 (17.7) | 140.3 (18.0)
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Test type: Non-Inferiority or Equivalence; p = 0.26, Mixed Models Analysis; Constrained longitudinal model adjusting for baseline stratification variables of diabetes status and blood pressure control; Mean Difference (Net) = -2.1, 95% CI 2-sided [-5.9 to 1.6]

3. Primary Outcome: Systolic Blood Pressure
Description: Continuous change in systolic blood pressure was measured as the primary outcome. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the12-month study visits.
Time Frame: 12 months
Population: Analysis Population Description: Analysis Population Description: 53 out of the 192 participants in the Titration Intervention group and 34 out of the 193 in the LPN control group had missing blood pressure measurement at 12 months due to not completing the assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 139 | 159
mmHg | 135.9 (15.7) | 138.4 (17.5)
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Test type: Non-Inferiority or Equivalence; p = 0.50, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.3, 95% CI 2-sided [-4.9 to 2.4]

4. Primary Outcome: Systolic Blood Pressure
Description: Continuous change in systolic blood pressure was measured as the primary outcome. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the18- month study visits.
Time Frame: 18 months
Population: 37 out of the 192 participants in the Titration Intervention group and 33 out of the 193 in the LPN control group had missing blood pressure measurement at 18 months due to not completing the assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 155 | 160
mmHg | 136.1 (17.6) | 138.0 (18.5)
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Test type: Non-Inferiority or Equivalence; p = 0.43, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Net) = -1.6, 95% CI 2-sided [-5.6 to 2.4]

5. Secondary Outcome: Number of Participants With Hypertension Control
Description: The investigators examined the difference in the degree of systolic BP control over the 18 months of the study between the intervention and control arms. Control was defined as SBP < 130mmHg for hypertensive patients with diabetes and < 140mmHg for patients without diabetes. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the baseline study visit.
Time Frame: Baseline
Population: Mean systolic blood pressure in control (units: participants)
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 192 | 193
Participants | 47 | 43

6. Secondary Outcome: Number of Participants With Hypertension Control
Description: The investigators examined the difference in the degree of systolic BP control over the 18 months of the study between the intervention and control arms. Control was defined as SBP < 130mmHg for hypertensive patients with diabetes and < 140mmHg for patients without diabetes. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the 6-month study visit.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 162 | 171
Participants | 66 | 63
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Comparison at 6 months; Test type: Non-Inferiority or Equivalence; p = 0.83, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link. Adjusted for baseline stratification variables of diabetes status; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.6]

7. Secondary Outcome: Number of Participants With Hypertension Control
Description: The investigators examined the difference in the degree of systolic BP control over the 18 months of the study between the intervention and control arms. Control was defined as SBP < 130mmHg for hypertensive patients with diabetes and < 140mmHg for patients without diabetes. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the 12-study visit.
Time Frame: 12 months
Population: 53 out of the 192 participants in the Titration Intervention group and 34 out of the 193 in the LPN control group had missing blood pressure measurement at 12 months due to not completing the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 139 | 159
Participants | 58 | 67
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Comparison at 12 months; Test type: Non-Inferiority or Equivalence; p = 0.53, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link. Adjusted for baseline stratification variables of diabetes status; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.5 to 1.4]

8. Secondary Outcome: Number of Participants With Hypertension Control
Description: The investigators examined the difference in the degree of systolic BP control over the 18 months of the study between the intervention and control arms. Control was defined as SBP < 130mmHg for hypertensive patients with diabetes and < 140mmHg for patients without diabetes. Mean systolic blood pressure was calculated by the average of 3 blood pressure measurements collected at the18- month study visit.
Time Frame: 18 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 155 | 160
Participants | 84 | 69
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Comparison at 18 months; Test type: Non-Inferiority or Equivalence; p = 0.09, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link. Adjusted for baseline stratification variables of diabetes status; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.9 to 2.3]

9. Secondary Outcome: Cost Effectiveness
Description: One of our secondary research questions was: "If the intervention results in greater reduction in SBP than the control group, is it cost effective?"
  Intervention results did not show statistically significant differences between arms, therefore cost effectiveness analysis was not appropriate.
  While cost effectiveness was not analyzed because it was a null trial, the investigators would have used resource utilization and cost data from VA data sets to measure VA outpatient and inpatient utilization and costs by arms over 18 months. The investigators would have examined hypertension-related outpatient pharmacy prescription counts and costs in order to compare them to total outpatient pharmacy costs and the investigators would have examined inpatient utilization and costs.
Time Frame: Over 18 months of study intervention
Population: Intervention results did not show statistically significant differences between arms, therefore cost effectiveness analysis is not appropriate.
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants Who Did Not Achieve Medication Adherence
Description: The investigators assessed adherence using patient self-report on a modified Morisky scale using 4 items:
  * Do you ever forget to take your blood pressure medicine?
  * Are you careless at times about taking your blood pressure medicine?
  * When you feel better do you sometimes stop taking you blood pressure medicine?
  * Sometimes if you feel worse when you take your blood pressure medicine, do you stop taking it? The scale is a Yes(0) or No (1) answer.
  A response of YES to any one of the 4 items indicated non-adherence, and responses of all no indicated adherence.
  The numbers in the descriptive tables reflect number non-adherent.
Time Frame: Baseline
Population: The numbers in the descriptive tables reflect #non-adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 192 | 193
Participants | 82 | 82

11. Secondary Outcome: Number of Participants Who Did Not Achieve Medication Adherence
Description: as for outcome 10
Time Frame: 6 months
Population: 30 out of the 192 participants in the Titration Intervention group and 21 out of the 193 in the LPN control group had missing medication adherence at 6 months due to not completing the assessment.
  The numbers in the descriptive tables reflect #non-adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 162 | 172
Participants | 62 | 69
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Test type: Non-Inferiority or Equivalence; p = 0.95, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link. Adjusted for baseline stratification variable of diabetes status and diabetes control; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.7 to 1.5]

12. Secondary Outcome: Number of Participants Who Did Not Achieve Medication Adherence
Description: as for outcome 10
Time Frame: 12 months
Population: 53 out of the 192 participants in the Titration Intervention group and 34 out of the 193 in the LPN control group had missing medication adherence at 12 months due to not completing the assessment.
  The numbers in the descriptive tables reflect #non-adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 139 | 159
Participants | 61 | 59
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Comparison at 12 months; Test type: Non-Inferiority or Equivalence; p = 0.12, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link.Adjusted for baseline stratification variable of diabetes status and blood pressure control; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.9 to 2.1]

13. Secondary Outcome: Number of Participants Who Did Not Achieve Medication Adherence
Description: as for outcome 10
Time Frame: 18 months
Population: 37 out of the 192 participants in the Titration Intervention group and 33 out of the 193 in the LPN control group had missing medication adherence at 18 months due to not completing the assessment.
  The numbers in the descriptive tables reflect #non-adherent.
Measure: Count of Participants; unit: Participants
Arm/Group | Titration Intervention | LPN Control
Number analyzed (Participants) | 155 | 160
Participants | 73 | 68
Statistical Analysis 1: Comparison: Titration Intervention vs LPN Control; Comparison at 18 months; Test type: Non-Inferiority or Equivalence; p = 0.30, Generalized Estimating Equation; Generalized Estimating Equation with a Logit Link. Adjusted for baseline stratification variables of diabetes status and blood pressure control; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.8 to 1.9]

ADVERSE EVENTS:
Time Frame: 18 months
Description: It is expected that these patients will have a variety of episodes related to cardiovascular and related diseases such as diabetes, age, smoking and drinking. These may include, but are not limited to, heart attack, stroke, and complications of diabetes among those patients with the disease, the diagnosis of cancer and dementia, development of disease of the lung or liver.
Arm/Group | Titration Intervention | LPN Control
All-Cause Mortality (participants affected / at risk) | 3/192 | 2/193
Serious Adverse Events (participants affected / at risk) | 40/192 | 9/193
Other Adverse Events (participants affected / at risk) | 117/192 | 112/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration Intervention (N=192) | LPN Control (N=193)
ER Visit (Renal and urinary disorders) | 0 (0) | 1 (1)
ER Visit (Infections and infestations) | 1 (1) | 1 (1)
ER Visit (Cardiac disorders) | 3 (4) | 0 (0)
ER Visit (Endocrine disorders) | 1 (1) | 0 (0)
Heart Attack (Cardiac disorders) | 3 (4) | 0 (0)
Hospitalization Other (Cardiac disorders) | 6 (7) | 3 (3)
Hospitalization Other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization Other (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hospitalization Other (General disorders) | 1 (1) | 0 (0)
Hospitalization Other (Infections and infestations) | 1 (1) | 1 (1)
Hospitalization Other (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hospitalization Other (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hospitalization Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hospitalization Other (Renal and urinary disorders) | 2 (3) | 0 (0)
Hospitalization Other (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hospitalization Other (Surgical and medical procedures) | 7 (10) | 0 (0)
Hospitalization Other (Vascular disorders) | 1 (1) | 0 (0)
Other (Cardiac disorders) | 1 (1) | 1 (1)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Other (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration Intervention (N=192) | LPN Control (N=193)
ER Visit (Cardiac disorders) | 13 (15) | 15 (25)
ER Visit (Gastrointestinal disorders) | 9 (9) | 6 (7)
ER Visit (General disorders) | 20 (24) | 22 (31)
ER Visit (Infections and infestations) | 17 (20) | 21 (31)
ER Visit (Injury, poisoning and procedural complications) | 13 (14) | 2 (2)
ER Visit (Musculoskeletal and connective tissue disorders) | 20 (31) | 26 (39)
ER Visit (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (12)
Hospitalization Other (Cardiac disorders) | 11 (11) | 11 (19)
Hospitalization Other (Surgical and medical procedures) | 11 (12) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT01390272/Prot_000.pdf
  • Informed Consent Form (2014-08-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT01390272/ICF_001.pdf